CLINICAL TRIAL: NCT01348217
Title: Prodige 26: Radiochemotherapy With and Without Dose Escalation in Patients Presenting Locally Advanced or Inoperable Carcinoma of the Oesophagus
Brief Title: Radiochemotherapy With and Without Dose Escalation in Patients Presenting Locally Advanced or Inoperable Carcinoma of the Oesophagus
Acronym: CONCORDE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Collaborators: National Cancer Institute, France (Other Government); UNICANCER (Other); SFRO:French Society of Radiation Oncology (Unknown); Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0291-1crgi09
Record Dates: First submitted 2011-04-29; First posted 2011-05-05 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Esophageal Cancer
Keywords: unoperated cancers; oesophagus; radiochemotherapy; with and without increased doses
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARM A (Active Comparator): Conformal 3D Radiotherapy with " ENI "-type prophylactic irradiation of the lymph nodes:
  1. Radiotherapy 40 Gy, in 20 fractions / 4 weeks: PTV (1cm in every direction)
  2. Boost 10 Gy in 5 fr: PTV = +1cm.
  3. Chemotherapy FOLFOX 4: 6 treatments in 3 courses concomitant to the radiotherapy (D1, D15, D29)
  Interventions: Radiation: Conformal 3D Radiotherapy with " ENI "-type prophylactic irradiation of the lymph node; Radiation: Boost; Drug: chemotherapy: FOLFOX 4
- ARM B (Experimental): Conformal 3D Radiotherapy with " ENI "-type prophylactic irradiation of the lymph nodes:
  1. 40 Gy in 20 fractions / 4 weeks, PTV (1cm in every direction)
  2. Boost 26 Gy in 13 fr: PTV = +1cm.
  3. Chemotherapy: FOLFOX 4: 6 treatments with 4 courses concomitant to radiotherapy (D1, D15, D29, D43).
  Interventions: Radiation: Conformal 3D Radiotherapy with " ENI "-type prophylactic irradiation of the lymph node; Radiation: Boost; Drug: chemotherapy: FOLFOX 4

INTERVENTIONS:
Radiation: Conformal 3D Radiotherapy with " ENI "-type prophylactic irradiation of the lymph node — 40 Gy in 20 fractions / 5 weeks, PTV (1cm in every direction)
Radiation: Boost — Boost 10 Gy in 5 fr, PTV = +1cm.
  Arms: ARM A
Radiation: Boost — Boost 26 Gy in 13 fr, PTV = +1cm.
  Arms: ARM B
Drug: chemotherapy: FOLFOX 4 — 6 treatments with 4 courses concomitant to radiotherapy (D1, D15, D29, D43) arm B or 3 courses concomitant to radiotherapy (D1, D15, D29) arm A.

SUMMARY:
Exclusive concomitant radiochemotherapy (RCT) at a dose of 50 Gy delivered over 5 weeks, according to the RTOG 85-01 protocol, has led to improved 5-year survival in 25% of patients, whereas no patients survived for 5 years using radiotherapy alone for patients with esophageal cancer. Surgery, even when combined with preoperative RCT, also gives disappointing results for locally advanced tumors, which casts serious doubts on the usefulness of preoperative radiotherapy. By varying the fractionation schedule, the length of treatment or the radiotherapy volumes, it has become possible to obtain levels of loco-regional relapse of around 35 to 45%. After reviewing the results for loco-regional relapse according to the dose of radiation and the recommended radiotherapy volumes, we aimed to investigate why increasing the dose of radiation has no impact in esophageal cancers. Although INT-0123 phase III trial showed no benefit of dose escalation in esophageal cancer, some issues remain unclear as most of the patients who died in the experimental arm were treated above 50Gy. Moreover, only the tumor was treated up to 64Gy while involved nodes were not considered for dose escalation in this trial. In the RTOG 85-01phase III trial, an elective nodal irradiation from subclavicular fossa up to the esophagogastric junction was performed with a 2D technique, delivering 30Gy which could be considered as not appropriate.

In this randomized phase II/III trial, we aim to test an exclusive concomitant chemoradiotherapy for patients with non resectable esophageal cancer with a dose escalation up to 66Gy on the primary tumor as well as the involved nodes using a 3D conformal technique combined with a 40 Gy elective nodal irradiation on lymph node stations (as defined by the RTOG) with a risk of microscopic involvement ≥ 20%.

ELIGIBILITY:
Inclusion Criteria:

1. Age> or = 18 and < 75 ans
2. WHO Status 0, 1 and 2
3. Enteral or parenteral feeding (> or = 1500 KCal) planned before the start of treatment
4. Histologically proven carcinoma of the oesophagus
5. Histological Types: adenocarcinomas and epidermoid carcinomas
6. T3, N0-N1-N2-N3, M0 (TNM version 7)
7. T1-T2, N0-N1-N2-N3, M0 with a contra-indication for surgery (TNM version 7)
8. Absence of trachea-oesophageal fistula
9. Written informed consent
10. Woman under appropriate contraception
11. Patient able to understand and complete, with help if necessary, a quality of life questionnaire

Exclusion Criteria:

1. Evolutive heart failure or myocardial necrosis for less than 6 months
2. Myocardial infarction of more than 6 months with ischemic sequelae on myocardial scintigraphy.
3. Patient cannot absorb at least 1500kcal/j before and/or during treatment
4. Left heart failure.
5. Stage II to IV arteriopathy in the Leriche and Fontaine classification
6. Creatinine > or = 1.25x N
7. PNN < 1,5.109 /l
8. Platelets < 100. 109 /l
9. Albumin < 30g/l
10. TP < 60% without anticoagulant
11. VEMS < 1l
12. History of cancer (except baso-cellular cutaneous epithelioma or in situ epithelioma of the cervix) that has relapsed in the 5 years preceding recruitment for the trial
13. Patient already enrolled in another therapeutic trial with an experimental molecule
14. Women who are pregnant or likely to be so, or who are breastfeeding
15. People who are in custody or under guardianship
16. Impossibility to adhere to the medical follow up for the trial for geographical,social or psychiatric reasons.
17. Presence of a history of radiotherapy to the chest or upper abdomen for another tumour
18. Peripheral neuropathy > or = grade 1 (CTC v3.0)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2011-05-06 (Actual); Primary Completion 2011-06-07 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Evaluate the rate of acute toxicity leading to cessation or temporary interruption of treatment of more than a total of 14 days or of 7 consecutive days during the whole treatment. | end of phase II (january 2014)
Evaluate the rate of completes endoscopic response at 3 months | for each patient 3 months after the end treatment
Survival without locoregional relapse at 2 years (time elapsed between date of randomisation and onset of local relapse and/or lymph node involvement) | after the end of phase III in january 2015 (anticipated)

SECONDARY OUTCOMES:
Evaluate adherence | every 3 months until the end of phase II (january 2014)
Evaluate acute toxicity at 3 months | for each patient 3 months after the end treatment
Evaluate death due to toxicity | each month during all the study
Evaluate quality of life (QLQ-C30 [annex n° 2] + OG25 [annex n° 3]) | after the completion of phase II (january 2014)
Compare according to treatment arm :Quality of life (QLQ-C30 [annex n° 2] + OG 25 [annex n° 3]) | after the completion of phase III (january 2015-anticpated)
Compare according to treatment arm :Overall survival | after the completion of phase III (january 2015-anticpated)
Compare according to treatment arm :Disease-free survival | after the completion of phase III (january 2015-anticpated)
Compare according to treatment arm :Acute and late toxicity according to the CTCAE version 3.0 scale | after the completion of phase III (january 2015-anticpated)
Compare according to treatment arm :The number of palliative interventions, the time to the first palliative intervention | after the completion of phase III (january 2015-anticpated)
Compare according to treatment arm :The rate of dysphagia according to Atkinson's criteria | after the completion of phase III (january 2015-anticipated)
Compare according to treatment arm :Survival without local recurrence in responders | after the completion of phase III (january 2015-anticipated)
Compare according to treatment arm :Progression-free survival in non-responding patients | after the completion of phase III (january 2015-anticipated)
Evaluation of the post-operative morbi-mortalities | after the completion of phase III (january 2015-anticipated)
  Evaluation of the post-operative morbi-mortalities (in 30 days) of the group of patients which will benefit from of a surgery of the tumoral residue.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Créhange, MD, Principal Investigator — Centre Georges Francois Leclerc
Locations (1):
- Centre Georges François Leclerc, Dijon, France

REFERENCES:
- [Derived] Bednarek C, Crehange G, Quivrin M, Cueff A, Vulquin N, Chevalier C, Cerda T, Petegnief Y, Mazoyer F, Maingon P, Bosset JF, Servagi Vernat S. Mapping of failures after radiochemotherapy in patients with non-metastatic esophageal cancer: A posteriori analysis of the dose distribution in the sites of loco-regional relapse. Radiother Oncol. 2015 Aug;116(2):252-6. doi: 10.1016/j.radonc.2015.07.019. Epub 2015 Jul 27. PMID 26228970